CLINICAL TRIAL: NCT07230041
Title: In Vivo Antibiotics Removal During Treatment With Hemoadsorption Cartridges and Continuous Renal Replacement Therapy in the Intensive Care Unit
Brief Title: In Vivo Antibiotics Removal During Hemoadsorption Cartridges and Continuous Renal Replacement Therapy in the Intensive Care Unit
Acronym: ICARO
Status: Recruiting | Type: Observational
Sponsor: Niguarda Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 4747
Record Dates: First submitted 2025-08-23; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Septic Shock
Keywords: antibiotic; target drug monitoring; meropenem; linezolid; daptomycin; in vivo
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICU patients with a diagnosis of infection/sepsis/septic shock: * stage 3 KDIGO consensus criteria, indication to CRRT
  * use of at least one of the following antibiotics meropenem, linezolid and daptomycin
  Interventions: Diagnostic Test: Liquid Chromatography - Tandem Mass Spectrometry

INTERVENTIONS:
Diagnostic Test: Liquid Chromatography - Tandem Mass Spectrometry — The samples will be processed by a company with expertise in antibiotic TDM. To ensure the highest standards of accuracy and reliability in our data, blood samples collected during this study will be evaluated using state-of-the-art Liquid Chromatography - Tandem Mass Spectrometry (LC-MS/MS) techniques. This advanced analytical method allows for the precise quantification and identification of biochemical compounds within complex biological matrices, providing unparalleled sensitivity and specificity. Following collection, blood is centrifuged to separate serum or plasma, which is then aliquoted to avoid degradation from freeze-thaw cycles. Aliquots are stored at -80°C to preserve sample integrity until analysis. This meticulous pre-analytical preparation ensures that all samples can be analyzed simultaneously, reducing analytical variability, and maintaining the quality of the samples for LC-MS/MS analysis

SUMMARY:
The purpose of this study is to measure the change in plasma concentrations of antibiotics used during passage through the CRRT filter and hemadsorption cartridge in patients with septic shock and renal failure requiring CRRT.

All patients aged > 18 years, admitted to the ICU, diagnosed with septic shock and renal failure requiring CRRT, receiving antibiotic therapy with at least one of the following drugs: meropenem, linezolid, and daptomycin, who provided informed consent, are included in the study.

Patients not admitted to the ICU, patients with renal failure not requiring CRRT, patients aged < 18 years, or those who did not provide informed consent are excluded. The enrollment period will last 12 months and will run from September 2024 to September 2025. The expected number of patients enrolled is twenty. To proceed with the study, after starting antibiotic therapy, a 4 ml dose of blood will be drawn (Vacuette tube ref. 454092) before the cartridge, immediately after, and after the dialysis filter. This measurement will be repeated after 4, 8, and 12 hours, which represents the maximum usage time of the cartridge.

After 12 hours, the cartridge becomes saturated and loses its adsorption capacity.

The CRRT filter, however, remains in place for at least 72 hours before being replaced. Treatment is maintained until clinically necessary.

For patients in intensive care, several blood samples are required throughout the day, both with a blood sample sent to the biochemistry laboratory every 6-8 hours to check clinical conditions, and with an arterial blood sample (blood gas) to check respiratory and metabolic status in patients on mechanical ventilation. Furthermore, in patients undergoing CRRT, electrolyte balance must be monitored every 4 hours. Therefore, the blood sample for the study inevitably coincides with one of the routine blood samples.

The test tube, labeled with a unique code, will be sent to the central laboratory, which will centrifuge the blood and extract the plasma. This aliquot will then be stored at -80°C in a dedicated space and sent to the designated laboratory upon analysis.

Determination of the plasma dosage of the antibiotic in use is commonly performed on patients admitted to the Intensive Care Unit, where clinically necessary. Participation in the study does not change current clinical practices.

DETAILED DESCRIPTION:
In ICU setting, most empiric antibiotic treatments include a combination of anti-Gram-positive and -negative bacteria, according to the different clinical scenarios. Thus, there are different possible regimen combinations, including two different drugs. We considered meropenem/linezolid (or daptomycin) as the drugs of choice in septic shock empiric treatment.

The motivation for the use of HA380 was to remove inflammatory cytokines. Only one HA 380 application (=12 hours) will be evaluated in this study.

Hemadsorption will be performed using a BBraun OMNI machine: a Jafron HA380 cartridge is assembled in series with a BBraun OMNI PLUS 'open' filter.

Hemadsorption lasts from 2 to 12 hours maximum, at the end the cartridge can be disassembled and CRRT treatment alone can be carried forward.

CRRT is performed according to the Omni machine BBraun protocol . CVVHD is the technique of choice because the diffusion method guarantees membrane stability.

A predilution Trisodium Citrate 4% infusion is performed, and filter anticoagulation is monitored via post filter blood samples with a target post filter ionized calcium (iCa+) values between 0,2- and 0,4 mmol/L. The citrate plasmatic starting dose is 4 mmol/L: the Omni machine automatically adjusts citrate flow in the predilution pump according to blood flow value, and vice versa. Post filter iCa+ values are checked 5 minutes after treatment institution and 5 minutes after every citrate's dose change; periodic checks are performed every 6 to 8 hours.

Blood flow varies according to patients' weight, dialysate to blood flow (expressed in ml/h) is kept constant in a 1:3 ratio, a table with reference values is provided by the manufacturer. A calcium free dialysate solution with an HCO3 concentration < 25 mmol/l is used.

A Calcium Chloride infusion is performed to restore a normal plasmatic iCa+ concentration. Calcium infusion takes place directly in the Omni circuit's venous line via a dedicated tubing. Starting calcium infusion dose is 1,7 mmol/l, patient's plasmatic iCa+ levels are checked before treatment's start, 30 minutes and 2 hours after treatment's start. Routine monitoring samples are performed every 6 to 8 hours.

When antibiotic treatment includes a loading dose, blood samples will be taken one hour after starting the continuous infusion.

Samples will be taken pre cartridge, post cartridge (pre filter) and after filter at baseline (at least 30 minutes after the beginning of CRRT treatment) and after 4-8 and 12 hours, according to the theoretical cartridge saturation time.

Samples will be processed at the same time, at the end of the recruitment time.

The samples will be processed by a company with expertise in antibiotic TDM. To ensure the highest standards of accuracy and reliability in our data, blood samples collected during this study will be evaluated using state-of-the-art Liquid Chromatography - Tandem Mass Spectrometry (LC-MS/MS) techniques. This advanced analytical method allows for the precise quantification and identification of biochemical compounds within complex biological matrices, providing unparalleled sensitivity and specificity. Following collection, blood is centrifuged to separate serum or plasma, which is then aliquoted to avoid degradation from freeze-thaw cycles. Aliquots are stored at -80°C to preserve sample integrity until analysis. This meticulous pre-analytical preparation ensures that all samples can be analyzed simultaneously, reducing analytical variability, and maintaining the quality of the samples for LC-MS/MS analysis.

Sample size calculation

To assess the variability in concentration levels in patients undergoing Continuous Renal Replacement Therapy (CRRT), a study will be conducted to compare the concentration levels in the blood before and after passing through the CRRT filter. Given the preliminary nature of this study and logistical limitations, the sample size will be set at 10 patients. This sample size is determined based on the ability to detect a clinically significant difference in concentrations of at least 12.53 units, with an assumed standard deviation of 10 units, while maintaining a significance level (α) of 0.05 and a study power (1-β) of 80%. This configuration ensures that the study has the capacity to identify significant differences of relevant magnitude, despite the relatively small number of participants. The decision to limit the sample size to 10 subjects reflects a balance between operational feasibility and the goal of obtaining valid and informative statistical results.

ELIGIBILITY:
Inclusion Criteria:

* stage 3 KDIGO consensus criteria, indication to CRRT
* use of at least one of the following antibiotics meropenem, linezolid and daptomycin
* < 18 yo

Exclusion Criteria:

* < 18 yo

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients with a diagnosis of infection/sepsis/septic shock
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
drug concentration | 4 hours
  assess the percentage of drug concentration variation pre and post HA 380 cartridge

SECONDARY OUTCOMES:
drug concentration variation | 8 and 12 hours
  assess the percentage of drug concentration variation pre and post HA 380 cartridge

CONTACTS AND LOCATIONS:
Overall Officials: Sara Micol Santambrogio, MD, Principal Investigator — Niguarda Hospital
Locations (1):
- Niguarda Hospital, Milan, Italia, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Not yet decided